CLINICAL TRIAL: NCT03332342
Title: Impact of Closed Eye Neutrophils on Dry Eye Disease Pathogenesis: Investigation on Repeatability and Effectiveness of an Eye Wash at Awakening for Diagnosis and Therapy
Brief Title: Closed Eye Neutrophils in Dry Eye Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Allergan Sales, LLC (Industry)
Responsible Party: Principal Investigator, Kelly Nichols, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 000517538
Record Dates: First submitted 2017-10-25; First posted 2017-11-06 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Dry Eye; Ocular Inflammation
Keywords: dry eye disease; tears; inflammation; ocular surface
MeSH Terms: conditions — Dry Eye Syndromes; Lacerations; Inflammation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Daily rinse of ocular surface (Experimental): Eye wash of the ocular surface with one teaspoon of saline immediately upon awakening, performed daily.
  Interventions: Other: Eye wash
- Weekly rinse of ocular surface (Active Comparator): Eye wash of the ocular surface with one teaspoon of saline immediately upon awakening, performed weekly.
  Interventions: Other: Eye wash
- Occasional rinse of ocular surface (Experimental): Eye wash of the ocular surface with one teaspoon of saline immediately upon awakening, performed on two separate occasions
  Interventions: Other: Eye wash

INTERVENTIONS:
Other: Eye wash — Research subjects will perform a wash of their ocular surface with phosphate buffered saline

SUMMARY:
The purpose of this prospective study is to evaluate different inflammatory cells that accumulate on the ocular surface, during sleep, and how these cells may contribute to dry eye disease. This study will involve at-home self-collection of tears using an eye wash method with sterile saline solution. While a diagnostic technique, the eye wash may also have a therapeutic benefit in dry eye sufferers, which will be assessed in the second phase of this project.

DETAILED DESCRIPTION:
Every night during sleep, there is an influx of white blood cells on to the surface of the eye. These cells likely perform a protective function, but it is also possible that their dysregulation could lead to disease. Using a larger cohort, our investigation hopes to better understand the function of these cells and their potential to be linked to dry eye disease. Further, the way in which these cells are collected, using an at-home self-collection of tears using an eye wash method with sterile saline solution, immediately upon awakening, could potentially provide relief to dry eye sufferers if performed on a daily basis.

ELIGIBILITY:
Inclusion Criteria:

* able to understand and sign an informed consent and HIPAA privacy document
* greater than 18 years of age at time of informed consent
* able and willing to follow protocol instructions, including performing at-home washes of the ocular surface and subsequent delivery of those samples to campus on a regular basis
* must be willing to have blood drawn

Exclusion Criteria:

* contact lens wear within past three months
* current consumption of cigarettes or tobacco, including e-cigarettes
* participation in any investigational drug studies within 30 days of informed consent
* pregnancy, by self-report
* active ocular infection or inflammation
* any refractive surgery within the past year
* any present Accutane (Isotretinoin) use
* any medication usage that, in the investigator's opinion, could be expected to interfere with the study, such as current use of topical steroids, Restasis, or Xiidra
* have any uncontrolled systemic disease, that in the investigator's opinion could be expected to interfere with the study, for example, conditions associated with dry eye disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2019-05-14 (Actual)

PRIMARY OUTCOMES:
Comfort assessment using the dry eye questionnaire | Baseline to 4 weeks
  Mean change from baseline in comfort following daily ocular surface washes
Comfort assessment using the ocular surface disease index | Baseline to 4 weeks
  Mean change from baseline in comfort following daily ocular surface washes

SECONDARY OUTCOMES:
Repeatability of diagnostic in measuring leukocyte count | Baseline to 4 weeks
  Repeatability of the eye wash in terms of leukocyte count, as measured by flow cytometry
Repeatability of diagnostic in measuring leukocyte phenotype | Baseline to 4 weeks
  Repeatability of the eye wash in terms of leukocyte phenotype, as measured by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Kelly K Nichols, OD MPH PhD, Principal Investigator — UAB School of Optometry
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No